CLINICAL TRIAL: NCT01631279
Title: A Phase I/II, Multi-Center, Open-Label, Dose Escalation Trial of the Safety and Pharmacokinetics of Intravenous PR610 Given Weekly in Subjects With Solid Tumors
Brief Title: A Dose Escalation Trial of PR610 Treating Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was prematurely discontinued due to unacceptable toxicity.
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR610-1001
Record Dates: First submitted 2012-06-07; First posted 2012-06-29 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: NSCLC; non-small cell lung cancer; non-squamous, non-small cell lung cancer; solid tumors; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PR610 (Experimental)
  Interventions: Drug: PR610

INTERVENTIONS:
Drug: PR610 — Dose escalation of PR610 to determine maximum tolerated dose for weekly administration

SUMMARY:
The purpose of this study is to determine the Maximum Tolerated Dose and the Dose-Limiting Toxicity of the drug to further evaluate safety and antitumor activity.

DETAILED DESCRIPTION:
Following informed consent, subjects undergo baseline evaluation and disease assessment. PR610 is administered intravenously weekly.

In the absence of progressive disease or unacceptable toxicity, subjects may continue to receive PR610. Intra-subject dose escalation (to no higher than the highest safe level) is allowed in subjects who are not experiencing dose limiting toxicity. Disease assessment will be repeated at week 6 and then every 8 weeks thereafter.

Pharmacokinetic (PK) assessment (PR610 and PR610E) will be performed for all subjects.

After determination of the MTD and the determination of the phase II dose, additional subjects with NSCLC that is genetically resistant to reversible EGFR inhibitors will be accrued into an expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 years or more
* Histologically-confirmed, progressive cancer with the following diagnosis:

  1. Phase I: locally advanced or metastatic solid tumor that may respond to an EGFR inhibitor;
  2. Phase II: Stage IIIB or IV, non-squamous, non-small cell lung cancer (NSCLC) with known sensitizing mutations in EGFR, and the T790M resistance mutation
* Failed, refused, or not eligible for standard of care therapy
* ECOG performance status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* At least 4 weeks from prior anticancer therapy including chemotherapy, hormonal, investigational, and/or biological therapies and irradiation. Ongoing hormonal therapy administered for control of prostate cancer which may be continued through the study. In addition, in the phase II portion of the study, prior reversible EGFR tyrosine kinase inhibitor therapy, such as erlotinib or gefitinib, may be continued up to 48 hours prior to start of PR610 to prevent significant disease flare.
* Recovered from prior treatment related toxicity

  1. except for grade 1 fatigue, grade 1 peripheral sensory neuropathy and grade 1 or 2 alopecia during the phase I portion of the study
  2. except for grade 1 toxicity, and grade 2 peripheral neuropathy during the phase II portion of the study
* At least four (4) weeks from prior major surgery
* Women of child-bearing potential must be willing to use an acceptable contraceptive method and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial
* Sexually active men must be willing to use an acceptable contraceptive method
* Adequate hematological and biological function
* Willingness to participate in PK sampling during cycles 1 and 2
* Willingness to provide permission to access archived tumor samples for evaluation of EGFR mutation status
* Willingness to provide samples for storage of normal tissue containing wild-type DNA

Additional Inclusion Criteria during Expansion Phase

* At least one target lesion as defined by RECIST 1.1 that allows for evaluation of tumor response

Exclusion Criteria:

* Pregnant or nursing women
* Any uncontrolled medical illness including, but not limited to, significant gastrointestinal disorders, cardiovascular disease, or interstitial lung disease
* History of clinically significant cardiovascular abnormalities, eg., uncontrolled hypertension, CHF (NYHA classification ≥2), unstable angina, poorly controlled arrhythmias, myocardial infarction within 6 months of study entry, implantable pacemaker or implantable cardioverter defibrillator
* Clinically significant abnormal 12-lead ECG with QTcF >450 msec
* Use of any medications known to produce QT prolongation
* Family history of Long QT Syndrome
* Prior treatment with anthracyclines with a cumulative dose of doxorubicin (or equivalent) ≥400 mg/m2
* Cardiac left ventricular function with resting ejection fraction of less than 50%
* Symptomatic CNS lesions or known CNS lesions that require therapy
* Prior history of an allergic reaction to a tyrosine kinase inhibitor

Additional Exclusion Criteria during Expansion Phase

* Any other malignancy likely to effect the assessment of toxicity or efficacy of PR610

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose (MTD) of PR610 for Both a 1-hour and a 24-hour Weekly IV Infusion | 3 weeks (1 cycle)
  The first cohort of three subjects will receive PR610 at Dose Level 1. Subsequent cohorts will receive PR610 at a dose levels determined as per dose escalation criteria. The MTD will be defined as the dose level at which one (1) or fewer subject in six exhibit DLT with the next highest dose level demonstrating two (2) or more of six (6) subjects with DLT (or for which more than ≥33% of subjects exhibit DLT if the cohort size exceeds 6 subjects).
Determine the Dose-Limiting Toxicity (DLT) of PR610 for Both a 1-hour and a 24-hour Weekly IV Infusion | 3 weeks (1 Cycle)
  DLT is defined as the following:
  * Occurs during the first cycle of PR610
  * Is considered PR610-related, as defined by "Definitely-related", "Probably-related" or "Possibly-related"
  * Is clinically significant, as determined by the Principal Investigator
  In addition, DLT will meet at least one of the criteria listed below using grading criteria from the CTCAEv4.
  * Grade 4 hematologic toxicity
  * Any drug-related toxicity that prevents administration of 100% of all doses of PR610 planned for Cycle 1
  * Grade 3 or higher non-hematologic toxicity

SECONDARY OUTCOMES:
Evaluate the safety profile of PR610: Adverse Events | 30 days following the last administration of study treatment
  The number of adverse events experienced by participants will be measured.
Peak Plasma Concentration (Cmax) of PR610 and PR610E for Both a 1-hour and a 24-hour Weekly Infusion | pre, 30 minutes into infusion, end of infusion, 1, 2, 4, 24, 48, and 72 hours post-infusion on Cycles 1 and 2
Evaluate the activity of PR610 in a general phase I population and in a subset of subjects with NSCLC genetically resistant to reversible EGFR inhibitors | 30 days following the last administration of study treatment
  Efficacy will be determined for each subject that received at least one dose of PR610 and had at least one post-baseline disease assessment. The following four outcomes will be tabulated:
  Tumor response Time to response Duration of response Progression-free survival
Time of Peak Plasma Concentration (tmax) of PR610 and PR610E for Both a 1-hour and a 24-hour Weekly Infusion | pre, 30 minutes into infusion, end of infusion, 1, 2, 4, 24, 48, and 72 hours post-infusion on Cycles 1 and 2
Half life (t1/2) of PR610 and PR610E for Both a 1-hour and a 24-hour Weekly Infusion | pre, 30 minutes into infusion, end of infusion, 1, 2, 4, 24, 48, and 72 hours post-infusion on Cycles 1 and 2
Area Under the Curve (AUC) of PR610 and PR610E for Both a 1-hour and a 24-hour Weekly Infusion | pre, 30 minutes into infusion, end of infusion, 1, 2, 4, 24, 48, and 72 hours post-infusion on Cycles 1 and 2
Clearance (CL) of PR610 and PR610E for Both a 1-hour and a 24-hour Weekly Infusion | pre, 30 minutes into infusion, end of infusion, 1, 2, 4, 24, 48, and 72 hours post-infusion on Cycles 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Proacta Inc., Study Chair — Proacta, Incorporated
Locations (6):
- United States (4):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - University of California-Davis Comprehensive Cancer Ctr, Sacramento, California
  - Robert H. Lurie Comprehensive Cancer Research Center, Chicago, Illinois
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Waikato